CLINICAL TRIAL: NCT06490224
Title: Can the Subjective Aspects of Health be Measured and Visually Displayed Without Harming Patient Experience: A Randomized Control Trial
Brief Title: Measuring and Displaying the Subjective
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PROM Prototyping
Record Dates: First submitted 2024-06-25; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Physician-Patient Relations; Communication Research

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Usual patient reported outcome measures
  Interventions: Behavioral: Relevant Patient Reported Outcome Measures (PROMs)
- Experimental (Experimental): Usual patient reported outcome measures + new visual display of responses to subjective health questions
  Interventions: Behavioral: Relevant Patient Reported Outcome Measures (PROMs); Other: My Whole Health Map

INTERVENTIONS:
Behavioral: Relevant Patient Reported Outcome Measures (PROMs) — Depending on the participant's complaint: Hip disability and osteoarthritis outcome score JR (HOOS JR), Knee disability and osteoarthritis outcome score JR (KOOS JR), Quick Disabilities of the Arm, Shoulder, and Hand, Quick Disabilities of the Arm, Shoulder, and Hand (QUICKDASH), Patient Health Questionnaire 9 (PHQ-9), General Anxiety Disorder-7 (GAD7), Patient Self-Efficacy Questionnaire (PSEQ-2), Patient-Reported Outcomes Measurement Information System (PROMIS Global 10)
Other: My Whole Health Map — Short visual map of responses to 10 questions of subjective measures.
  Arms: Experimental

SUMMARY:
The investigators developed a brief set of subjective health measures designed to feel more relevant to patients seeking musculoskeletal specialty care, presented the scores to patients and clinicians using an easy-to-understand visual display, and measured whether or not this process harmed patient experience.

DETAILED DESCRIPTION:
Musculoskeletal patient-reported outcome measures (PROMs; measures of levels of discomfort and incapability) were originally designed as tools for clinical research as were other self-reported measures of the subjective aspects of illness such as mental health measures. PROMs and mental health measures are increasingly used in clinical practice with individual patients. A few areas for improvement are noted in the use of questionnaires in musculoskeletal specialty care, including relevancy, understandability, and their confusing use in heath strategies. The investigators sought to assess the impact of an enhanced and more personalized self-reported health measurement strategy to address some of these opportunities by developing a brief set of items addressing levels of discomfort, incapability, mental, and social health designed to feel relevant to musculoskeletal specialty care and resulting in an easy-to-understand display that can be a communication tool for patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* All new and return patients
* English and Spanish speakers

Exclusion Criteria:

* Cognitive deficiency precluding PROM completion
* Language other than English or Spanish

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
CollaboRATE survey | Immediately after the intervention
  Quality of shared decision-making (Numerical scale from 1-27; Higher scores equal better outcome)
Jefferson Scale Patient Perceptions of Physician Empathy (JSPPPE) | Immediately after the intervention
  Patient perceived clinician empathy (Numerical scale from 1-35; Higher scores equal better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Jayakumar, MD. PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neil W. Wagle MM (2017) Implementing Patient-Reported Outcome Measures. NEJM Catal
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Amini M, Oemrawsingh A, Verweij LM, Lingsma HF, Hazelzet JA, Eijkenaar F, van Leeuwen N. Facilitators and barriers for implementing patient-reported outcome measures in clinical care: An academic center's initial experience. Health Policy. 2021 Sep;125(9):1247-1255. doi: 10.1016/j.healthpol.2021.07.001. Epub 2021 Jul 8. PMID 34311981